CLINICAL TRIAL: NCT02330029
Title: A Randomized, Double-blind, and Placebo-controlled Study on the Treatments of Irritable Bowel Syndrome
Brief Title: Pinaverium and Herbs for Irritable Bowel Syndrome Treatment: an Onset and Offset Study (PHIBEST)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Macrohard Institute of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D00320141210
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome,; Pinaverium; Herbal medication for IBS,; Tong Xie Yao Fang (Formula for pain and diarrhea)
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — pinaverium; diterpenoid C, Radix curcumae

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TCM (Traditional Chinese medicine) (Active Comparator): Formula for pain and diarrhea, Atractylodes (~10-15g), Paeonia Lactiflora (~15-30g), Tangerine Peel (~10g), Ledebouriella Root (~10g), Radix codonopsitis (~10-15g), Radix curcumae (~10g), Fingered citron (~10g), Tuckahoe (~15g), etc.
  Interventions: Device: Atractylodes; Device: Paeonia Lactiflora; Device: Tangerine Peel; Drug: Ledebouriella Root; Drug: Radix codonopsitis; Drug: Radix curcumae; Drug: Fingered citron; Drug: Tuckahoe
- Pinaverium (Active Comparator)
  Interventions: Drug: Pinaverium
- Placebo (Placebo Comparator): Placebo is blindly given to patients
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pinaverium — To test the effectiveness and safety of the formula for pain and diarrhea, we will randomly assign patients into one 3 groups: Pinaverium, TCM (Formula for pain and diarrhea) group, and placebo group, and treat them accordingly.
  Arms: Pinaverium
Device: Atractylodes — Atractylodes (~10-15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Device: Paeonia Lactiflora — Paeonia Lactiflora (~15-30g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Device: Tangerine Peel — Tangerine Peel (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Ledebouriella Root — Ledebouriella Root (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Radix codonopsitis — Radix codonopsitis (~10-15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Radix curcumae — Radix curcumae (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Fingered citron — Fingered citron (~10g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Tuckahoe — Tuckahoe (15g)
  Other Names: One of active ingredients in TCM group
  Arms: TCM (Traditional Chinese medicine)
Drug: Placebo — Placebo is blindly given to patients.
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the onset of action, offset of action, efficacy, and safety of pinaverium and an herbal medication for irritable bowel syndrome (IBS) for a long term (over one year). Pinaverium has been in many countries, but there is no randomized, double-blind, large sample size, and placebo-controlled study on this medication yet. Tong Xie Yao Fang (Formula for pain and diarrhea) is a historically and contemporarily used traditional Chinese medicine that can be used for IBS. The hypothesis is that the two remedies are effective and safe for IBS treatment with no significant different onset and offset of actions when tested by modern clinical standards and criteria.

DETAILED DESCRIPTION:
Pinaverium bromide (pinaverium), an antispasmodics, is one of the most commonly used IBS medication worldwide. However, original clinical studies on pinaverium are scarce. Only five original clinical studies from Europe, one from Latin America, and one from Asian were found. These studies were single-centered and small sample sized (19 - 53 IBS patients) studies.

Tong Xie Yao Fang has long been used in China. Its efficacy and safety has not been evaluated by modern scientific method.

Effectiveness, onset and offset of actions are the most considered factors when physicians choose medications for IBS. Yet, to our knowledge, there are no clinical studies studied the onset and offset of actions of pinaverium, which remains one of the most transcribed IBS medications, and herbs, which are becoming more popular for treating IBS.

This study is designed to evaluate onset and offset of actions, efficacy, and safety over a long term (>1 year) of pinaverium and Tong Xie Yao Fang for IBS treatment in a double-blind, randomized, and large sample size clinical trial using placebo as a control.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years old age group, male and female
* In accordance with the above Western medicine Rome III standards.
* In accordance with the above description of Deficient Spleen Qi and Liver Qi Stagnation
* Informed consent for treatment
* No change in appetite during treatments periods

Exclusion Criteria:

* Pregnant or lactation female patients, and Fertility male patients
* Present digestive system disease within current three months
* Take IBS medicines within ten days prior to treatment or during treatment
* Take depression medicine within ten days prior to treatment or during treatment
* Take pain reliever medicine within ten days prior to treatment or during treatment
* Have serious primary heart, liver, kidney, lung and blood system diseases, asthma, and Lung and liver dysfunction patients
* If an emergency occurs; a physician terminates the treatment
* Cannot comply with the rules and cannot cooperate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-11 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain | 2 years
  0 = no pain, 10 worst pain
Primary endpoint --- vi) Form (appearance) of stool | 2 years
  Use Bristol stool scale.

SECONDARY OUTCOMES:
Frequency of the pain | 2 year
  0 = no pain; 1 = 1 pain/day; 2 = 2 pains/day; 3 = 3 pains/day; ................... 9 = 9 pains/day; 10 = ≥ 10 pains/day.
# of stools per day | 2 years
  0 = no stool; 1 = 1 stool/day; 2 = 2 stools/day; 3 = 3 stools/day; ............... 9 = 9 stools/day; 10 = ≥ 10 stools/day.
Abdominal discomfort | 2 years
  0 = no discomfort...... 10 = Worst possible, unbearable unbearable discomfort
Frequency of discomfort | 2 years
  0 = no discomfort; 1 = 1 discomfort/day; 2 = 2 discomforts/day; 3 = 3 discomforts /day; ................... 9 = 9 discomforts/day; 10 = ≥ 10 discomforts/day.

OTHER OUTCOMES:
IBS global symptom relief | 2 years
  IBS global symptom relief was evaluated by each patient at the end of the therapy as "improved", "stayed the same", or "worsened"
Treatment-emergent adverse effect (TEAE) profiles. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Baiwen Li, MD, Principal Investigator — Department of Gastroenterology, Shanghai First People's Hospital, Shanghai Jiao Tong University, 100 Haining Rd. Hongkou, Shanghai 200280, China.
Locations (4):
- China (4):
  - Second Jiangsu Provincial Hospital of Traditional Chinese Medicine affiliated to Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial Hospital of Traditional Chinese Medicine affiliated to Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Beijing Xuanwu Hospital of Traditional Chinese Medicine affiliated to Capital Medical University., Beijing
  - Shanghai First People's Hospital affiliated to Shanghai Tiao Tong University, Shanghai

REFERENCES:
- [Derived] Zheng L, Lu W, Xiao Q, Lai Y, Fan H, Sun Y, Huang D, Wang Y, Li Z, Jiang Z, Liu X, Zhang L, Zuo D, Shou Z, Tang Q, Huang H, Yang Y, Tang Z, Xiao J. Assessing the post-treatment therapeutic effect of pinaverium in irritable bowel syndrome: a randomized controlled trial. Sci Rep. 2021 Jul 6;11(1):13894. doi: 10.1038/s41598-021-92990-7. PMID 34230526